CLINICAL TRIAL: NCT06575270
Title: Pulse Oximetry Accuracy and Skin Pigmentation in Congenital Heart Disease: A Prospective Observational Study
Brief Title: Skin Pigment/Pulse Oximeter in Congenital Heart Disease (CHD)
Status: Recruiting | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Garrett Burnett, Associate Professor, Icahn School of Medicine at Mount Sinai
Other Study IDs: STUDY-23-00956; TE00003017 (Other Grant/Funding Number: Anesthesia Patient Safety Foundation)
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-11

CONDITIONS: Hypoxemia; Skin Pigment; Congenital Heart Disease
Keywords: Pulse Oximetry; Skin Pigment; Congenital Heart Disease; Hypoxemia
MeSH Terms: conditions — Hypoxia; Pigmentation Disorders; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Pediatric Patients with Congenital Heart Disease: No intervention will take place in this observational study. All patients will have their skin pigment measured using a color spectrophotometer and color matching techniques (Fitzpatrick Scale, Monk Skin Tone Scale). Two pulse oximeters will be utilized and pulse oximeter readings will be compared to simultaneous measured arterial saturations. After cardiopulmonary bypass is initiated for the surgery, the subject's involvement in the study will be completed.

SUMMARY:
Recent retrospective studies have demonstrated differences between pulse oximeter values (SpO2) and measured arterial oxygen saturation (SaO2) in patients identifying as Black or Hispanic. These retrospective studies have limitations because self-reported race is likely not an accurate metric for level of skin pigmentation and the retrospective nature of these studies may impact the accuracy of simultaneous measures of arterial oxygen saturation and pulse oximeter values. The few prospective studies that have evaluated this issue have utilized color-matching techniques to quantify skin pigmentation, and fewer studies have directly measured skin pigmentation in relation it to pulse oximeter accuracy. The aim of this study is to prospectively measure pulse oximeter accuracy in relation to measured levels of skin pigmentation in the congenital heart disease population.

DETAILED DESCRIPTION:
This is a prospective observational study aiming to evaluate the relationship between pulse oximeter accuracy to the measured level of skin pigmentation in pediatric patients with congenital heart disease (CHD). These patients live with varying levels of hypoxemia, making them an ideal study population to investigate this critical patient safety issue. The study population will be pediatric patients (age <18 years old) with a diagnosis of congenital heart disease presenting for cardiac surgery at the Mount Sinai Hospital. These patient's will undergo surgery as per protocol, as if they were not in a research study, but will have their skin pigment measured using a non-invasive device (color spectrophotometer) prior to surgery. As part of the normal surgery protocols, arterial blood gas samples will be completed. The measured oxygen levels (SaO2) on arterial blood gas will be compared to the pulse oximeter value using simultaneous measurements to ensure the measures are concurrent. After cardiopulmonary bypass is initiated for the surgery, the subject's involvement in the study will be completed.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients (age less than 18 years old) with a diagnosis of CHD (cyanotic or acyanotic) who are presenting for cardiac surgery under general anesthesia with planned arterial access.

Exclusion Criteria:

* Age greater than 18 years old
* Emergency surgery
* Significant preoperative anemia (hemoglobin <8.0 g/dL)
* Preoperative hemodynamic instability (i.e., >1 vasoactive infusions or mechanical circulatory support)
* The presence of any colored nail polish on the planned site of pulse oximeter placement, planned use of any intravenous dyes intraoperatively, and patient, parent, or guardian refusal.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with a past medical history of congenital heart disease presenting for cardiac surgery under general anesthesia with anticipated arterial vascular access.
Sampling Method: Non-Probability Sample
Enrollment: 92 (Estimated)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Level of Skin Pigmentation | Day 1 of study participation
  Pulse oximeter accuracy as it relates to level of skin pigmentation as measured by color spectrophotometry. Pulse oximeter accuracy will be measured using the Accuracy Root Mean Squared (ARMS), mean bias, and proportional bias (Bland-Altman).

SECONDARY OUTCOMES:
Fitzpatrick Skin Tone Scale | Day 1 of study participation
  Pulse Oximeter Accuracy in measuring skin pigmentation as measured by Fitzpatrick Skin Tone Scale Pulse oximeter accuracy as it relates to level of skin pigmentation as measured by Fitzpatrick Scale. Scale from I-VI, with higher number indicating darker skin tone
Monk Skin Tone Scale | Day 1 of study participation
  Pulse oximeter accuracy as it relates to level of skin pigmentation as measured by Monk Skin Tone Scale. Scale from 1-10, higher numbers indicates darker skin tone.
Number of participants who experience at least one episode of occult hypoxemia | Day 1 of study participation
  Incidence of occult hypoxemia, defined as SpO2 ≥92% despite SaO2≤88%, as it relates to measured skin pigment and incidence of occult hypoxemia will be described. Incidence will be measured by assessing the total number of participants who experience at least one episode of occult hypoxemia.

CONTACTS AND LOCATIONS:
Overall Officials: Garrett W. Burnett, M.D., Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai Hospital, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon study completion and in accordance with any peer-reviewed journal requirements.
Access Criteria: Researchers who provide a methodologically sound proposal. To achieve aims in the approved proposal. Proposals should be directed to garrett.burnett@mountsinai.org. To gain access, data requestors will need to sign a data access agreement.